CLINICAL TRIAL: NCT04914702
Title: Continuous Monitoring of Vital Signs With Different Wearable Devices in Pediatric Patients Undergoing Chemotherapy for Cancer - a Comparison and Feasibility Pilot Study
Brief Title: Feasibility and Comparison of Continuously Monitored Vital Signs in Pediatric Patients With Cancer.
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: Bern/Basel 2021 WD Pilot
Record Dates: First submitted 2021-06-03; First posted 2021-06-07 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Pediatric Cancer; Febrile Neutropenia; Oncology; Chemotherapy-induced Neutropenia
Keywords: Wearable device; Everion®; CORE®; Continuous recording; Vital signs; Pediatric oncology
MeSH Terms: conditions — Neoplasms; Febrile Neutropenia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Everion® only: Two Everion® devices, one for the day and one for the night, to be switched every morning and evening, will be given to the participants for the duration of 2 weeks (fourteen days) with the instruction to wear all the time, with exception of the time needed for the patients' hygiene.
  Interventions: Device: Everion®
- CORE® only: A CORE® device will be given to the participants for the duration of 2 weeks (fourteen days) with the instruction to wear it all the time, with exception of the time needed for battery charging and the patients' hygiene.
  Interventions: Device: CORE®
- Everion® first, CORE® second: Two Everion® devices, one for the day and one for the night, to be switched every morning and evening, will be given to the participants for the duration of 2 weeks (fourteen days) with the instruction to wear all the time, with exception of the time needed for the patients' hygiene.
  Then a CORE® device will be given to the participants for the duration of 2 weeks (fourteen days) with the instruction to wear it all the time, with exception of the time needed for battery charging and the patients' hygiene.
  Interventions: Device: Everion®; Device: CORE®
- CORE® first, Everion® second: A CORE® device will be given to the participants for the duration of 2 weeks (fourteen days) with the instruction to wear it all the time, with exception of the time needed for battery charging and the patients' hygiene.
  Then two Everion® devices, one for the day and one for the night, to be switched every morning and evening, will be given to the participants for the duration of 2 weeks (fourteen days) with the instruction to wear all the time, with exception of the time needed for the patients' hygiene.
  Interventions: Device: Everion®; Device: CORE®
- Everion® and CORE® simultaneously: Two Everion® devices, one for the day and one for the night, to be switched every morning and evening, and one CORE® will be given to the participants for the duration of 2 weeks (fourteen days) with the instruction to wear all the time, with exception of the time needed for the patients' hygiene.
  Interventions: Device: Everion®; Device: CORE®

INTERVENTIONS:
Device: Everion® — The Everion® is an on-skin wearable devices measuring vital signs. It will be given to the participants for the duration of 2 weeks (fourteen days) with the instruction to wear all the time, with exception of the time needed for the patients' hygiene.
  Groups: CORE® first, Everion® second; Everion® and CORE® simultaneously; Everion® first, CORE® second; Everion® only
Device: CORE® — The CORE® is an on-skin wearable devices measuring vital signs. It will be given to the participants for the duration of 2 weeks (fourteen days) with the instruction to wear all the time, with exception of the time needed for the patients' hygiene.
  Groups: CORE® first, Everion® second; CORE® only; Everion® and CORE® simultaneously; Everion® first, CORE® second

SUMMARY:
In this pilot study the feasibility continous recording of vital signs in pediatric patients under chemotherapy for cancer, is studied.

Vital signs and are recorded with two different wearable devices (WDs): Everion®, by Biovotion (now Biofourmis), Zurich, Switzerland and CORE® by GreenTEG, Zurich, Switzerland. Patients can choose if they want to wear one or both WDs during this study. Those opting to wear two WDs can choose if they want to wear them in parallel, or sequentially.

Results from the two different WDs will be compared. Study duration for each participant is 14 days per device.

DETAILED DESCRIPTION:
In a previous study (Bern 2019 WD Pilot, NcT04134429) the investigators found that continuous recording of vital signs with the Everion® is feasible in good quality across a wide age range (3 to 16 years) of pediatric patients undergoing chemotherapy for cancer. However, the pre-defined criterion to claim feasibility was not formally reached and low compliance was the main reason identified.

In this study the investigators want to assess the impact of measures aiming to increase compliance on feasibility for the Everion®.

Second, the investigators want to assess the feasibility of a second device, made commercially available only in October 2020, the CORE® WD by GreenTEG. Results from the two different wearable devices will be compared. Study duration for each participant is 14 days per device.

ELIGIBILITY:
Inclusion Criteria:

* Chemotherapy treatment because of any malignancy, expected to last ≥1 month at time of recruitment for myelosuppressive therapy; or at least one cycle of myeloablative therapy requiring autologous (Bern/Basel) or allogeneic (Basel) hematopoietic stem cell transplantation.
* Age from 1 month to 17.99 years at time of recruitment
* Written informed consent from parents and participants, where applicable

Exclusion Criteria:

* Local skin diseases prohibiting wearing of the WD.
* Denied written informed consent from participants

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients undergoing chemotherapy for cancer treated in the departments of pediatric oncology at the Children's university hosptials Bern or Basel.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of continous recording of core temperature with the two wearable devices (WDs) | 14 days
  The primary outcome is defined as at least sufficient data quality (Everion® ≥50, quality score 0 (lowest) to 100 (best); CORE® ≥2, quality score 1 (lowest) to 4 (best)) of core temperature measurement, with arrival on dashboard ≤30 minutes after recording, during a cumulative duration of ≥18/24h per day (midnight to midnight), on ≥7 days within the 14 days of the study period.

SECONDARY OUTCOMES:
Feasibility of continous recording of heart rate with the Everion® | 14 days
  At least sufficient data quality (Everion® ≥50, quality score 0 (lowest) to 100 (best) of heart rate measurement, with arrival on dashboard ≤30 minutes after recording, during a cumulative duration of ≥18/24h per day (midnight to midnight), on ≥7 days within the 14 days of the study period.
Feasibility of continous recording of heart rate variability with the Everion® | 14 days
  At least sufficient data quality (Everion® ≥50, quality score 0 (lowest) to 100 (best) of heart rate variability measurement, with arrival on dashboard ≤30 minutes after recording, during a cumulative duration of ≥18/24h per day (midnight to midnight), on ≥7 days within the 14 days of the study period.
Feasibility of continous recording of respiration rate with the Everion® | 14 days
  At least sufficient data quality (Everion® ≥50, quality score 0 (lowest) to 100 (best) of respiration rate measurement, with arrival on dashboard ≤30 minutes after recording, during a cumulative duration of ≥18/24h per day (midnight to midnight), on ≥7 days within the 14 days of the study period.
Cumulative time of monitoring core temperature with the two wearable devices (WDs) | 14 days
  Cumulative length of time with recorded core temperature with at least sufficient data quality (Everion® ≥50, quality score 0 (lowest) to 100 (best); CORE® ≥2, quality score 1 (lowest) to 4 (best)) per study day.
Cumulative time of monitoring heart rate with the Everion® | 14 days
  Cumulative length of time with recorded heart rate with at least sufficient data quality (Everion® ≥50, quality score 0 (lowest) to 100 (best)) per study day.
Cumulative time of monitoring heart rate variability with the Everion® | 14 days
  Cumulative length of time with recorded heart rate variability with at least sufficient data quality (Everion® ≥50, quality score 0 (lowest) to 100 (best)) per study day.
Cumulative time of monitoring respiration rate with the Everion® | 14 days
  Cumulative length of time with recorded respiration rate with at least sufficient data quality (Everion® ≥50, quality score 0 (lowest) to 100 (best)) per study day.
Data arrival on the dashboard for core temperature (Everion®) | 14 days
  Cumulative length of time with data arrival on the dashboard ≤30 minutes after recording (continuous outcome, measured daily) for core temperature for the Everion®
Data arrival on the dashboard for core temperature (CORE®) | 14 days
  Cumulative length of time with data arrival on the dashboard ≤30 minutes after recording (continuous outcome, measured daily) for core temperature for the CORE®
Effort for investigators assessed by number of contacts | 14 days
  Cumulative number of contacts with the participants for the Investigators.
Effort for investigators assessed by duration of contacts | 14 days
  Cumulative duration of contacts with the participants for the Investigators.
Acceptability of Everion® | 14 days
  Proportion of participants indicating that continuous monitoring with the Everion® is acceptable (binary outcome, measured once).
Acceptability of CORE® | 14 days
  Proportion of participants indicating that continuous monitoring with the CORE® is acceptable (binary outcome, measured once).
Side Effects | 14 days
  Number and description of side effects reported by participants, if applicable (categorical outcome) and comparison of the side-effects of the two different WDs.
User-friendliness | 14 days
  Comparison of the user-friendliness and preference of the different WDs as judged by the participants (categorical outcome, assessed with questionnaires)
Comparison of core temperature with discrete measurements | 14 days
  Difference between discrete measurements of core temperature, performed by the participants, if applicable, twice daily or more if clinically indicated and the measured signal from both WDs at the corresponding time.
Exploration | 14 days
  Exploration of potential changes in or specific patterns of all measured signals within 48 hours before clinical diagnosis of fever, with or without neutropenia, if applicable.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Brack, MD, PhD, Principal Investigator — Pediatric Hematology/Oncology, Inselspital, Bern University Hospital; Christa Koenig, MD, Study Chair — Pediatric Hematology/Oncology, Inselspital, Bern University Hospital
Locations (2):
- Switzerland (2):
  - University Children's Hospital Basel, University of Basel, Basel
  - Inselspital, Bern

IPD SHARING:
Plan to Share IPD: Yes
The coded study data (from the WD and clinical data) will be uploaded to figshare and made publically available for other researchers.
Supporting Information: Study Protocol
Time Frame: After publication of the study results, no time limitation after publication.
Access Criteria: Open Access

REFERENCES:
- [Derived] Koenig C, Ammann RA, Schneider C, Wyss J, Roessler J, Brack E. Continuous timely monitoring of core temperature with two wearable devices in pediatric patients undergoing chemotherapy for cancer - a comparison study. Support Care Cancer. 2024 Feb 24;32(3):188. doi: 10.1007/s00520-024-08366-w. PMID 38400942